CLINICAL TRIAL: NCT03439852
Title: Increasing Physical Activity in Filipino Lay Leaders
Brief Title: Modifying Physical Activity and Sedentary Time in Filipino Faith Leaders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R15MD011474 (NIH)
Record Dates: First submitted 2018-02-07; First posted 2018-02-20 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Physical Activity and Sedentary Behavior; Healthy Aging
Keywords: physical activity; Sedentary time
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: cluster randomized controlled trial comparing physical activity/sedentary time intervention to delayed treatment condition
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators blinded to outcome follow-up data reported by study condition until completion of intervention period. Outcomes assessor blinded to participant identity - data entered only with ID number
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light to Moderate Physical Activity/Sedentary behavior (Experimental): The telephone counseling plus group cohesion intervention is designed to increase Light-to-Moderate intensity physical activity (LMPA) and reduce Sedentary time (ST). The 12-wk intervention includes group discussions during 3 regular monthly club meetings when clubs' accumulated milestones for LMPA/ST min/wk will be identified and future cumulative club goals for PA/ST set. In addition, each member will receive 12 weekly personalized phone calls from health coaches who will use motivational interviewing to set individualized LMPA/ST goals setting, reduce barriers, and facilitate social support for LMPA/ST change.
  Interventions: Behavioral: Light-to-Moderate Physical Activity / Sedentary Time
- Delayed Treatment/Healthy Aging (No Intervention): Delayed Treatment (DT) / Healthy Aging materials Condition is for 12 weeks and participants receive 12 phone calls using a previously developed contact-matched protocol that uses mailed healthy aging information and telephone calls to assess symptom ratings. After the initial 12 weeks they then receive the LMPA/ST intervention

INTERVENTIONS:
Behavioral: Light-to-Moderate Physical Activity / Sedentary Time — 12 weeks of telephone counseling -motivational interviewing designed to increase leisure-time physical activity and decrease amount of sitting each day
  Other Names: LMPA/ST
  Arms: Light to Moderate Physical Activity/Sedentary behavior

SUMMARY:
The outcomes of this application will provide nursing researchers with information about ways to increase physical activity (PA) and decrease sedentary time (ST) in at-risk older Filipinos adults who are lay leaders in Filipino Catholic clubs in Hawaii. The proposed 12-week PA/ST program will include both a group-based component (3 group discussions during monthly club meetings) and a personalized telephone counseling component (12 weekly calls from nursing students to problem solve barriers to increasing light-to-moderate physical activity and decreasing / breaking up sedentary time). The project will stimulate multidisciplinary research at our School of Nursing and School of Medicine and has the potential to help older at-risk Filipinos reach national guidelines for healthy levels of physical activity and lower the amount of time they spend sitting/being sedentary.

DETAILED DESCRIPTION:
Asian-Americans (A-As) are under-represented in chronic disease research, including lifestyle interventions. A-As are 42% of population in Hawaii and across the U.S. they are projected to more than double to 34.4 million by 2060, with a much higher proportion of older A-As compared to other races. Within A-As, Filipino-Americans have high rates of hypertension, diabetes, and chronic kidney disease, especially as they age. This is largely due to unhealthy diets, high BMIs, sedentary behaviors, and low physical activity (PA). Our previous work found Filipino seniors are under-active and spend > 8 hours a day in sedentary time (ST). About 90% of Filipinos in Hawaii are Catholic and previous PA interventions involving faith-based organizations have been shown to be culturally relevant for ethnic minorities and can effectively increase PA. Our innovative application focuses on changing both PA and ST in 250 Filipino lay leaders who represent their parish within the Oahu Council of Filipino Catholic Clubs (OCFCCs). OCFCCs maintain Filipinos' Catholic traditions and their cultural heritage. This project builds on our previous research with Filipino leaders from these clubs, and our expertise with effective PA and ST interventions. Team includes 3 nursing faculty, 1 medical school faculty, a project director, and from 9-12 graduate /undergraduate nursing students. The students will participate in a community-engaged 3-yr research project relevant both to their future research efforts and their use of self-management strategies with patients who at-risk for chronic diseases. The investigators will develop, implement, and test the efficacy of a culturally tailored PA/ST intervention for under-active/sedentary Filipino seniors (ages: 55-75 yrs) some of who may have multiple morbidities under medical control. The investigators will initially strengthen our partnership with OCFCC by engaging council members in semi-structured meetings where key cultural and familial issues that hinder/facilitate PA/ST will be discussed, the project's name/logo will be created, and plans to facilitate clubs' engagement across 3-year project will be solidified. Specific Aims: 1) test the efficacy of a Light-to-Moderate PA-LMPA/ST intervention with ten OCFCC clubs (25 lay leaders/club; n = 250 total) that will be randomly assigned to either a 12wk LMPA/ST intervention consisting of 3 group discussions during club meetings plus 12 counseling calls, or to Delayed Treatment condition initially given health education materials and 12 contact-matched calls on topics unrelated to PA/ST; then, the LMPA/ST intervention. 2) test maintenance of LMPA/ST 12 wks after LMPA/ST intervention ends. 3) analyze LMPA/ST self-report & accelerometer data collected at baseline, 12, 24, and 36 wks, and test demographic, psychosocial, environmental, and group factors as mediators/moderators of change in LMPA/ST. 4) discuss project findings with statewide Diocesan Congress of Filipino Catholic Clubs and the feasibility of using lay leaders to change the LMPA/ST of their parishioners from churches across Hawaii via a train-the-trainer lay leader model. This project will stimulate community engaged/team science research at our School of Nursing and enhance students' research skills.

ELIGIBILITY:
Inclusion Criteria:

* Member in one of 10 Filipino Catholic Clubs (within the Oahu Council of Filipino Catholic Clubs) on the island of Oahu in the state of Hawaii

Exclusion Criteria:

1. Age: less than 55 years OR older than 75 years of age
2. Planning to move (off the island of Oahu) in the next 9 months
3. Body Mass Index: If BMI is < 18.5 or > 40 (we will be measuring their height and weight to determine BMI at enrollment)
4. Currently exercising: Regularly (weekly) active at a moderate intensity* or higher >60 minutes a week (* = brisk walk)
5. Currently in Treatment: Actively having cancer treatment or in physical therapy following surgery/stroke
6. A recent (in last 6 months) diagnosis of: Cancer, Heart disease, had a heart attack, Lung disease, Chronic Kidney Disease, Stroke, or underwent surgery
7. Physician recommends that person have only supervised physical activity (i.e., in a health care / physical therapy setting)
8. Needs a cane or walker (or other assistive device) to walk especially outdoors on uneven surfaces

Need health care provider's approval/clearance before enrollment if potential participant has the following:

1. Asthma or other respiratory disease made worse by exercise
2. A heart valve problem or is taking medications for a heart condition
3. Severe osteoarthritis
4. Insulin dependent Type 1 or Type 2 diabetes (or often has a blood glucose > 235 mg/dl or 13mmol/L) (need MD clearance if do not know blood glucose)
5. Diagnosis/Treatment for Cancer over last 12 months or had a Stroke in the past (> 6 months ago)
6. Resting blood pressure ≥ 160/90 (with or without medications) (need MD clearance if do not know BP)
7. Has chest pain when exercising or recently (last 4 weeks) developed any chest pain (i.e., when not doing physical activity)
8. Has tendency to lose consciousness or collapse from dizziness
9. Has a bone or joint problem that could be aggravated by physical activity

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clementina Ceria-Ulep, PhD, Principal Investigator — University of Hawaii; Cheryl L Albright, PhD, Principal Investigator — University of Hawaii
Locations (1):
- University of Hawaii at Manoa, Office of Research Services, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be available for Univ. of Hawaii graduate students/post-doctoral fellows who have been involved in the project for dissertations or publications, first, then to others. Individuals wishing to use our data will be required to fill out a Data Sharing Request Form, which asks for information on the type of data set being requested, anticipated data use, research questions, study design, variables, analysis plan, and human subjects approval. We will also plan for general release and sharing of deidentified data (following the acceptance for publication of the main findings from the study) as we believe this to be essential for expedited translation of research results into larger arenas to improve human health.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred onsite at Catholic churches in the community.
Pre-assignment Details: If the participants' self reported height/weight (i.e, BMI) (collected anonymously to determine eligibility prior to signing a consent form) was below our BMI cutpoint, but their measured height and weight exceeded our BMI cutpoint (measured after consent form signed), participants were excluded from study before condition-specific information was provided.
Groups:
- Light to Moderate Physical Activity/Sedentary Time: The telephone counseling plus group cohesion intervention is designed to increase Light-to-Moderate intensity physical activity (LMPA) and reduce Sedentary time (ST). The 12-wk intervention includes group discussions during 3 regular monthly club meetings when clubs' accumulated milestones for LMPA/ST min/wk will be identified and future cumulative club goals for PA/ST set. In addition, each member will receive 12 weekly personalized phone calls from health coaches who will use motivational interviewing to set individualized LMPA/ST goals setting, reduce barriers, and facilitate social support for LMPA/ST change.
  Light-to-Moderate Physical Activity / Sedentary Time: 12 weeks of telephone counseling -motivational interviewing designed to increase leisure-time physical activity and decrease amount of sitting each day
Period: Baseline to 12 Weeks
Arm/Group | Light to Moderate Physical Activity/Sedentary Time | Delayed Treatment/Healthy Aging
Started (baseline enrollment) | 12 | 23
Completed (Completed 12 wk survey) | 8 | 16
Not Completed | 4 | 7
Not completed — Failed complete 12 wk survey | 4 | 7
Period: 12weeks to 24weeks
Arm/Group | Light to Moderate Physical Activity/Sedentary Time | Delayed Treatment/Healthy Aging
Started | 8 | 16
Completed | 6 | 16
Not Completed | 2 | 0
Not completed — failed complete 12 or 24 wk surveys | 2 | 0
Period: 24 Weeks to 36 Weeks Follow up
Arm/Group | Light to Moderate Physical Activity/Sedentary Time | Delayed Treatment/Healthy Aging
Started | 6 | 16
Completed | 5 | 16
Not Completed | 1 | 0
Not completed — failed to complete 36 wk survey | 1 | 0

BASELINE CHARACTERISTICS:
Population: Adults recruited from community-based Catholic Churches
Groups:
- Total: Total of all reporting groups
Arm/Group | Light to Moderate Physical Activity/Sedentary Time | Delayed Treatment/Healthy Aging | Total
Number analyzed (Participants) | 12 | 23 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] — Collected via baseline survey
  years | 65.5 (6.6) | 63.8 (6.1) | 64.4 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 18 | 28
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 22 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — All participants were recruited from Hawaii
  participants
    United States | 12 | 23 | 35
Minutes per week physical activity [Mean (Standard Deviation); unit: minutes per week] — minutes per week (light-to moderate intensity)
  minutes per week | 180 (207) | 171 (175) | 174 (183)
Minutes/week of High-Light physical activity [Mean (Standard Deviation); unit: minutes per week] — CHAMPS questionnaire measure of "High-Light" physical activity (i.e, activities with MET values between 2 and 3
  minutes per week | 445 (274) | 335 (300) | 370 (293)
Breaks per hour at baseline [Mean (Standard Deviation); unit: breaks per hour] — number of breaks per hour when sitting at home
  breaks per hour | 2.5 (1.7) | 1.1 (1.0) | 1.8 (1.3)
Sitting time hours per day [Mean (Standard Deviation); unit: hours per day] | 5.4 (4.9) | 6.3 (6.3) | 5.8 (5.6)
Breaks per hour in sitting time at work [Mean (Standard Deviation); unit: breaks per hour] — The Workplace Sitting Breaks Questionnaire (SITBRQ) asked respondents to consider the past 7 days, and report how many breaks from sitting were taken in an hour at work and at home. This could include standing, stretching, or taking a short walk. Participants were asked to not count lunch breaks/coffee breaks at work (or breaks to prepare meals at home).
  breaks per hour | 2.6 (1.8) | 1.5 (1.5) | 2.05 (1.65)

OUTCOME MEASURES:

1. Primary Outcome: Minutes Per Week of Hi/Light Intensity Physical Activity
Description: The Community Health Activities Model Program for Seniors (CHAMPS) survey was used to assess this outcome. Participants reported the number of times/week they do a specific physical activity, and then choose one of 6 time frames that represent the amount of time they did that activity, from less than one hr/week to 9 or more hours/week. Minutes per week of high-light intensity were defined as the sum of all the minutes of physical activities with >2 and <3 Metabolic Equivalents (METs).
Time Frame: Measured at Baseline and after 12 weeks
Population: Analyses were performed on randomized participants who provided both a baseline and 12-week (follow-up) assessment (survey), regardless of the level of physical activity/sedentary time they reported during a phone call, the number of condition-specific telephone calls they received, or the number of LMPA/ST condition group cohesion sessions they attended. Four participants in LMPA/ST condition and 7 participants in DT/HG condition did not provide a 12-week assessment.
Measure: Mean (Standard Deviation); unit: minutes per week
Groups:
- Light-to-Moderate Physical Activity and Sedentary TIme Condition: The telephone counseling plus group cohesion intervention was designed to increase Light-to-Moderate intensity physical activity (LMPA) and reduce Sedentary Time (ST). The 12-wk intervention includes group discussions during 3 regular monthly club meetings when clubs' accumulated milestones for LMPA/ST min/wk were identified and future cumulative club goals for PA/ST set. In addition, each member received 12 weekly phone calls from health coaches who used motivational interviewing to set individualized LMPA/ST goals setting, reduce barriers, and facilitate social support for LMPA/ST change.
- Delayed Treatment/Healthy Aging Condition: Delayed Treatment (DT) / Healthy Aging materials Condition lasted for 12 weeks and participants received 12 phone calls using a previously developed contact-matched protocol that used mailed healthy aging information and telephone calls to assess daily symptom ratings. After the initial 12 weeks they then received the LMPA/ST intervention
Arm/Group | Light-to-Moderate Physical Activity and Sedentary TIme Condition | Delayed Treatment/Healthy Aging Condition
Number analyzed (Participants) | 11 | 23
minutes per week
  Baseline | 445 (274) | 335 (300)
  12 weeks: number analyzed (Participants) | 7 | 16
  12 weeks | 626 (271) | 493 (330)
Statistical Analysis 1: Comparison: Light-to-Moderate Physical Activity and Sedentary TIme Condition vs Delayed Treatment/Healthy Aging Condition; Multilevel modeling for repeated measures was conducted to compare 2 conditions over time. The model included group, time, and the interaction between group and time, adjusting for within-subject correlation. The response was transformed using squared root to satisfy the model assumption; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = 0.83, 95% CI 2-sided [0.26 to 1.39]

2. Primary Outcome: Minutes Per Week of Moderate-to-vigorous Intensity Physical Activity
Description: The CHAMPS survey was used to assess this outcome. Minutes per week of moderate-to-vigorous intensity physical activity were defined as the sum of all the minutes of physical activities with >3 METs. For both conditions this was from baseline to at 12 weeks
Time Frame: Measured at Baseline and after 12 weeks
Population: Analyses on participants who provided a pre and post intervention survey, regardless of the level of physical activity/sedentary time they reported during a phone call, the number of condition-specific telephone calls they received, or the number of LMPA/ST group cohesion sessions they attended. Four participants in LMPA/ST condition and 7 participants in DT/HG condition did not provide a 12-week assessment.
Measure: Mean (Standard Deviation); unit: minutes per week
Groups:
- Light to Moderate Physical Activity/Sedentary Behavior Condition: The telephone counseling plus group cohesion intervention is designed to increase Light-to-Moderate intensity physical activity (LMPA) and reduce Sedentary time (ST). The 12-wk intervention includes group discussions during 3 regular monthly club meetings when clubs' accumulated milestones for LMPA/ST min/wk will be identified and future cumulative club goals for PA/ST set. In addition, each member will receive 12 weekly personalized phone calls from health coaches who will use motivational interviewing to set individualized LMPA/ST goals setting, reduce barriers, and facilitate social support for LMPA/ST change.
  Light-to-Moderate Physical Activity / Sedentary Time: 12 weeks of telephone counseling -motivational interviewing designed to increase leisure-time physical activity and decrease amount of sitting each day
- Delayed Treatment/Healthy Aging Condition: Delayed Treatment (DT) / Healthy Aging materials Condition is for 12 weeks and participants receive 12 phone calls using a previously developed contact-matched protocol that uses mailed healthy aging information and telephone calls to assess symptom ratings. After the initial 12 weeks they then receive the LMPA/ST intervention
Arm/Group | Light to Moderate Physical Activity/Sedentary Behavior Condition | Delayed Treatment/Healthy Aging Condition
Number analyzed (Participants) | 11 | 23
minutes per week
  baseline | 180 (207) | 171 (175)
  12-weeks: number analyzed (Participants) | 7 | 16
  12-weeks | 238 (191) | 308 (268)
Statistical Analysis 1: Comparison: Light to Moderate Physical Activity/Sedentary Behavior Condition vs Delayed Treatment/Healthy Aging Condition; Multilevel modeling conducted for repeated measures comparing minutes per week of light-to-moderate physical activity for participants in two conditions over time. In the multilevel models, participants were nested within Catholic Clubs, adjusting for within-club and within-subject correlations. The model includes group, time, and the interaction between group and time, adjusting for within-subject correlation. The response was transformed using squared root to satisfy the model assumption; Test type: Superiority; p = 0.05, Mixed Models Analysis — Calculated; Median Difference (Net) = 1.14, 95% CI 2-sided [-0.37 to 2.64]

3. Primary Outcome: Minutes Per Week Hi/Light Intensity Physical Activity
Description: The CHAMPS survey was used to assess this outcome. Participants reported the number of times/week they do a specific physical activity, and then choose one of 6 time frames that represent the amount of time they did that activity, from less than one hr/week to 9 or more hours/week. Minutes per week of high-light intensity were defined as the sum of all the minutes of physical activities with >2 and <3 METs. For LMPA/ST condition, their post-intervention was at 12 weeks and their maintenance was at 24 weeks. For DT/HA condition, their post-intervention was at 24 weeks and their maintenance was at 36 weeks.
Time Frame: 12 weeks after LMPA intervention ended
Population: Analyses on participants who provided a 12 wk maintenance ( 12 wks after intervention ended) survey, regardless of the level of physical activity/sedentary time they reported during a phone call, the number of condition-specific telephone calls they received, or the number of LMPA/ST condition group cohesion sessions attended. Six participants in LMPA/ST condition and 6 in DT/HA condition did not provide a 24-week survey. At 36 weeks, 6 in DT/HA did not provide a survey
Measure: Mean (Standard Deviation); unit: Minutes per week
Arm/Group | Light to Moderate Physical Activity/Sedentary Behavior Condition | Delayed Treatment/Healthy Aging Condition
Number analyzed (Participants) | 6 | 17
Minutes per week
  Post-intervention | 626 (271) | 504 (430)
  Maintenance | 695 (408) | 550 (461)
Statistical Analysis 1: Comparison: Light to Moderate Physical Activity/Sedentary Behavior Condition vs Delayed Treatment/Healthy Aging Condition; Multilevel modeling for the repeated measures was conducted comparing the two conditions over time. In the multilevel models, participants were nested within Catholic Clubs, adjusting for within-club and within-subject correlations. The model includes group, time, and the interaction between group and time, adjusting for within-subject correlation. The response was transformed using squared root to satisfy the model assumption; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Net) = -0.72, 95% CI 2-sided [-2.31 to 0.88]

4. Secondary Outcome: Hours Per Week of Sedentary Time
Description: Sedentary behavior was measured via the Measure of Older Adults' Sedentary Time (MOST), a validated survey with good test-retest reliability and results from ST interventions have found it sensitive to change. The survey asked respondents to report the time they spent doing 7 different tasks/activities (over last week) while sitting or lying (other than sleeping/napping/ill in bed) including: (1) TV or video/DVD watching, (2) other screen use/internet use: computer/tablet/Smartphone, (3) reading, (4) socializing with friends or family (in-person or when talking on phone), (5) driving/riding in car or city bus, (6) doing hobbies, and (7) any other activities. The total time spent sitting for each task/activity and total across all tasks was calculated.
Time Frame: Baseline and after 12 weeks
Population: Table reports data from surveys collected at baseline and 12 weeks and the results from repeated measures analyses for hours per week of sedentary time
Measure: Mean (Standard Deviation); unit: Hours per week
Groups:
- Light to Moderate Physical Activity/Sedentary Time Condition: The telephone counseling plus group cohesion intervention is designed to increase Light-to-Moderate intensity physical activity (LMPA) and reduce Sedentary time (ST). The 12-wk intervention includes group discussions during 3 regular monthly club meetings when clubs' accumulated milestones for LMPA/ST min/wk will be identified and future cumulative club goals for PA/ST set. In addition, each member will receive 12 weekly personalized phone calls from health coaches who will use motivational interviewing to set individualized LMPA/ST goals setting, reduce barriers, and facilitate social support for LMPA/ST change.
  Light-to-Moderate Physical Activity / Sedentary Time: 12 weeks of telephone counseling -motivational interviewing designed to increase leisure-time physical activity and decrease amount of sitting each day
Arm/Group | Light to Moderate Physical Activity/Sedentary Time Condition | Delayed Treatment/Healthy Aging Condition
Number analyzed (Participants) | 12 | 23
Hours per week
  Baseline | 5.4 (4.9) | 6.3 (6.3)
  12 Weeks: number analyzed (Participants) | 8 | 16
  12 Weeks | 5.4 (3.9) | 6.5 (5.1)
Statistical Analysis 1: Comparison: Light to Moderate Physical Activity/Sedentary Time Condition vs Delayed Treatment/Healthy Aging Condition; Multilevel modeling for the repeated measures was conducted comparing the two conditions over time. In the multilevel models, participants were nested within Catholic Clubs, adjusting for within-club and within-subject correlations. The model includes group, time, and the interaction between group and time, adjusting for within-subject correlation; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = 0.96, 95% CI 2-sided [-2.67 to 4.60]

5. Secondary Outcome: Breaks in Sitting Time Per Hour at Home
Description: The Workplace Sitting Breaks Questionnaire (SITBRQ) asked respondents to consider the past 7 days, and report how many breaks from sitting were taken in an hour at work and at home. This could include standing, stretching, or taking a short walk. Participants were asked to not count breaks to prepare meals at home
Time Frame: baseline and after 12 weeks
Population: Participants were sent 3 surveys after baseline, at 12wk, 24wk, and 36 wks, if a participant did not complete one of these surveys he/she was still sent the next survey unless they had asked to be dropped from study
Measure: Mean (Standard Deviation); unit: breaks per hour
Arm/Group | Light to Moderate Physical Activity/Sedentary Time Condition | Delayed Treatment/Healthy Aging Condition
Number analyzed (Participants) | 12 | 23
breaks per hour
  baseline | 2.5 (1.7) | 1.1 (1.0)
  12 weeks: number analyzed (Participants) | 8 | 16
  12 weeks | 4.6 (1.5) | 1.7 (1.4)
Statistical Analysis 1: Comparison: Light to Moderate Physical Activity/Sedentary Time Condition vs Delayed Treatment/Healthy Aging Condition; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -0.76, 95% CI 2-sided [-1.11 to -0.40]

6. Secondary Outcome: Breaks Per Hour in Sitting Time at Work
Description: The Workplace Sitting Breaks Questionnaire (SITBRQ) asked respondents to consider the past 7 days, and report how many breaks from sitting were taken in an hour at work. This could include standing, stretching, or taking a short walk. Participants were asked to not count lunch breaks/coffee breaks at work
Time Frame: baseline and after 12 weeks
Population: number ofbreaks in sitting time at work
Measure: Mean (Standard Deviation); unit: breaks per hour in sitting at work
Arm/Group | Light to Moderate Physical Activity/Sedentary Time Condition | Delayed Treatment/Healthy Aging Condition
Number analyzed (Participants) | 12 | 23
breaks per hour in sitting at work
  baseline | 2.6 (1.8) | 1.5 (1.5)
  12 weeks: number analyzed (Participants) | 8 | 16
  12 weeks | 4.2 (1.3) | 1.4 (1.7)
Statistical Analysis 1: Comparison: Light to Moderate Physical Activity/Sedentary Time Condition vs Delayed Treatment/Healthy Aging Condition; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = -0.62, 95% CI 2-sided [-1.15 to 0.10]

7. Secondary Outcome: Percent That Met 150 Minutes of Moderate-to-vigorous Physical Activity (MVPA) Per Week
Description: Outcome was a binary variable reporting whether a participant met 150 min per week of MVPA at each of the two time points (1=met the recommendation, 0=did not meet).
Time Frame: baseline and after 12 weeks
Population: Participants were sent 3 surveys following baseline each 12 weeks apart (thus baseline, 12wk, 24wk, and 36wk). Some people did not complete one or more of the follow-up surveys. They were sent a survey at each time points unless they told us they no longer wanted to participate in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Light to Moderate Physical Activity/Sedentary Time Condition | Delayed Treatment/Healthy Aging Condition
Number analyzed (Participants) | 12 | 23
Participants
  baseline met 150 min MVPA: number analyzed (Participants) | 11 | 23
  baseline met 150 min MVPA | 6 | 9
  12-wks met 150 min MVPA: number analyzed (Participants) | 7 | 16
  12-wks met 150 min MVPA | 5 | 10
Statistical Analysis 1: Comparison: Light to Moderate Physical Activity/Sedentary Time Condition vs Delayed Treatment/Healthy Aging Condition; Test type: Superiority; p < 0.05, Mixed Models Analysis; Repeated measures generalized linear model test effects of time/group, & interaction rate met MVPA, adjusting for within subject correlation; Median Difference (Net) = -0.49, 95% CI 2-sided [-2.10 to 1.11]

ADVERSE EVENTS:
Time Frame: Continuous systematic collection adverse events after enrollment first began March, 2018 via surveys (collected 12, 24, 36 weeks after enrollment) and verbal questions at the end of telephone calls held weekly after enrollment for first 12 -24 weeks depending on condition.
Description: reported to study staff by participant on intervention phone call
Arm/Group | Light to Moderate Physical Activity/Sedentary Time | Delayed Treatment/Healthy Aging
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/23
Other Adverse Events (participants affected / at risk) | 0/12 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light to Moderate Physical Activity/Sedentary Time (N=12) | Delayed Treatment/Healthy Aging (N=23)
Serious adverse event - hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1) — Participant's appendix was removed, reported to DSMB who ruled unrelated to study interventions, reported to IRB also ruled not related to study interventions

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT03439852/Prot_SAP_002.pdf
  • Informed Consent Form (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/52/NCT03439852/ICF_003.pdf